CLINICAL TRIAL: NCT02892565
Title: Hypercoagulable Phenotype by Thrombinography (in Presence of C Protein Dynamic Inhibitory System): Marker of Venous Thrombosis Risk in Systemic Lupus and Antiphospholipid Syndrome? Case-control Study
Brief Title: Hypercoagulable Phenotype by Thrombinography (in Presence of C Protein Dynamic Inhibitory System)
Acronym: TACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: PHRC 2005/TACT-LECOMPTE/NK
Record Dates: First submitted 2016-09-02; First posted 2016-09-08 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Venous Thrombosis
Keywords: systemic lupus erythematosus; antiphospholipid syndrome; antiphospholipid antibodies
MeSH Terms: conditions — Venous Thrombosis; Lupus Erythematosus, Systemic; Antiphospholipid Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cases (Experimental): Patients with SLE and/or APL and first vein thrombosis episode
  Interventions: Other: Blood sample
- Controls (Other): age-matched; Patients with SLE and/or APL
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample

SUMMARY:
The purpose is to determine the hypercoagulable phenotype by thrombinography associated to an increased risk of symptomatic and objectively confirmed first venous thrombotic event. This is a case-control study in a population with patients having systemic lupus erythematosus (SLE) and/or antiphospholipid antibodies (APL).

Secondary purposes are:

1. To determine the frequency of hypercoagulable phenotype in study population;
2. To analyze the sensibility: consequences of variation of hypercoagulable phenotype threshold on the importance of risk;
3. To identify (genetic and not) factors for hypercoagulable phenotype and their frequency in different groups.

ELIGIBILITY:
Inclusion Criteria:

Cases :

* Patients with SLE and/or APL and first documented deep vein thrombosis episode (minimum 6 months, maximum 6 years)
* Any weight and height
* Absence of current anticoagulant treatment but possibility of platelet function inhibitory treatment; actual guidelines suggest long-term anticoagulant treatment in patients with first episode of venous thrombosis and having APL; however, these patients can be studied if they are in one of these circumstances: 1/ "inconvenient" stop by patient, 2/ aspirin decided by doctor after prolonged treatment

Controls:

* Patients with SLE and/or APL without thrombosis (venous or arterial)
* Any weight and height
* Possibility of platelet function inhibitory treatment (primary prophylaxis of arterial manifestations)

Exclusion Criteria:

Cases and Controls :

* Pregnancy
* Refusal of consent
* Difficulty of follow-up (not sufficient motivation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2005-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Thrombin potential measured with thrombinography | baseline
Measurement of IC50-APC (concentration of APC diminishing 50% thrombin potential at APC concentration = 0) | baseline

IPD SHARING:
Plan to Share IPD: No